CLINICAL TRIAL: NCT03016975
Title: Annular ReduCtion for Transcatheter Treatment of Insufficient Mitral ValvE (ACTIVE): A Prospective, Multicenter, Randomized, Controlled Pivotal Trial to Assess Transcatheter Mitral Valve Repair With Edwards Cardioband System and GDMT vs GDMT Alone in Patients With FMR and Heart Failure
Brief Title: Edwards Cardioband System ACTIVE Pivotal Clinical Trial (ACTIVE)
Acronym: ACTIVE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Procedure and device development
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-05
Record Dates: First submitted 2017-01-08; First posted 2017-01-11 (Estimated); Results first posted 2022-11-09 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Functional Mitral Regurgitation; Mitral Regurgitation; Mitral Insufficiency
Keywords: Edwards Cardioband; Mitral Valve; Transcatheter; Mitral repair; Functional mitral regurgitation; Secondary mitral regurgitation; Annuloplasty
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Randomized - Edwards Cardioband System (Experimental): Transcatheter mitral valve repair with the Edwards Cardioband System plus guideline directed medical therapy (GDMT)
  Interventions: Device: Edwards Cardioband System; Drug: Guideline Directed Medical Therapy
- Randomized - Control (Active Comparator): Guideline directed medical therapy (GDMT)
  Interventions: Drug: Guideline Directed Medical Therapy
- Roll-In - Edwards Cardioband System (Experimental): Transcatheter mitral valve repair with the Edwards Cardioband System plus guideline directed medical therapy (GDMT)
  Interventions: Device: Edwards Cardioband System; Drug: Guideline Directed Medical Therapy

INTERVENTIONS:
Device: Edwards Cardioband System — Transcatheter mitral valve repair with the Edwards Cardioband System
  Other Names: Transcatheter mitral valve repair (TMVr)
  Arms: Randomized - Edwards Cardioband System; Roll-In - Edwards Cardioband System
Drug: Guideline Directed Medical Therapy — GDMT Only

SUMMARY:
To establish the safety and effectiveness of the Edwards Cardioband System in patients with functional mitral regurgitation (FMR).

DETAILED DESCRIPTION:
The ACTIVE Trial is a prospective, randomized, multicenter trial. Patients with clinically significant functional mitral regurgitation will be randomized 2:1 to receive either transcatheter mitral valve repair with the Edwards Cardioband System plus guideline directed medical therapy (GDMT) or GDMT alone. Patients will be seen for follow-up visits at discharge, 30 days, 6 months, and annually through 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Clinically Significant Functional Mitral Regurgitation (MR);
* Symptomatic heart failure;
* Patient hospitalized due to heart failure during 12 months prior to submission to Central Screening Committee OR elevated Brain Natriuretic Peptid (BNP);
* Patient is able and willing to give informed consent and follow protocol procedures, and comply with follow-up visit compliance.

Exclusion Criteria:

* Primarily degenerative MR;
* Mitral annular calcification that would impede implantation of device;
* Other severe valve disorders requiring intervention;
* Mitral valve anatomy which may preclude proper Edwards Cardioband deployment;
* Life expectancy of less than twelve months;
* Patient is participating in concomitant research studies of investigational products which have not reached their primary endpoint;
* Unwillingness or inability to undergo follow-up investigations/visits;
* Other medical, social, or psychological conditions that precludes appropriate consent and follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2022-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Whisenant, MD, Principal Investigator — Intermountain Medical Center; Vinod Thourani, MD, Principal Investigator — Piedmont Heart Institute
Locations (24):
- United States (24):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of Colorado Denver, Aurora, Colorado
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - St. Vincent Heart Center, Indianapolis, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Morristown Medical Center, Morristown, New Jersey
  - NYU Langone Health, New York, New York
  - Columbia University Medical Center/New York Presbyterian Hospital, New York, New York
  - Lenox Hill Hospital - Northwell Health, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Sanger Heart & Vascular Institute - Atrium Health, Charlotte, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Providence Health &Services, Heart & Vascular Institute, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Pinnacle Health, Harrisburg, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia Health System, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Roll-in: Transcatheter mitral valve repair with the Edwards Cardioband System plus guideline directed medical therapy (GDMT). This patient group is treated by physicians requiring additional training prior to beginning randomized cohort enrollment.
- Experimental: Edwards Cardioband System: Transcatheter mitral valve repair with the Edwards Cardioband System plus guideline directed medical therapy (GDMT)
- Control: No Intervention: Guideline directed medical therapy (GDMT)
Period: At 30 Days Follow-up
Arm/Group | Roll-in | Experimental: Edwards Cardioband System | Control: No Intervention
Started | 12 | 0 | 0
Completed | 11 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Subject is a Screen failure | 1 | 0 | 0
Period: At 6 Months Follow-up
Arm/Group | Roll-in | Experimental: Edwards Cardioband System | Control: No Intervention
Started | 11 | 0 | 0
Completed | 6 | 0 | 0
Not Completed | 5 | 0 | 0
Not completed — Death | 2 | 0 | 0
Not completed — Subject withdrawn by investigator | 1 | 0 | 0
Not completed — Re-attempt procedure | 1 | 0 | 0
Not completed — Aborted implant | 1 | 0 | 0
Period: At 1 Year Follow-up
Arm/Group | Roll-in | Experimental: Edwards Cardioband System | Control: No Intervention
Started | 6 | 0 | 0
Completed | 6 | 0 | 0
Not Completed | 0 | 0 | 0
Period: At 2 Year Follow-up
Arm/Group | Roll-in | Experimental: Edwards Cardioband System | Control: No Intervention
Started | 6 | 0 | 0
Completed | 5 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0
Period: At 3 Year Follow-up
Arm/Group | Roll-in | Experimental: Edwards Cardioband System | Control: No Intervention
Started | 5 | 0 | 0
Completed | 3 | 0 | 0
Not Completed | 2 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: At 4-year Follow-up
Arm/Group | Roll-in | Experimental: Edwards Cardioband System | Control: No Intervention
Started | 3 | 0 | 0
Completed | 2 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Exited Study for other reasons | 1 | 0 | 0
Period: At 5-year Follow-up
Arm/Group | Roll-in | Experimental: Edwards Cardioband System | Control: No Intervention
Started | 2 | 0 | 0
Completed | 2 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data were not collected for the experimental or control group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Roll-in | Experimental: Edwards Cardioband System | Control: No Intervention | Total
Number analyzed (Participants) | 12 | 0 | 0 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.8 (9.60) |  |  | 71.8 (9.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  |  | 2
  Male | 10 |  |  | 10
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data unavailable for 3 patients
  Participants
    number analyzed (Participants) | 9 | 0 | 0 | 9
    American Indian or Alaska Native | 0 |  |  | 0
    Asian | 0 |  |  | 0
    Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
    Black or African American | 1 |  |  | 1
    White | 8 |  |  | 8
    More than one race | 0 |  |  | 0
    Unknown or Not Reported | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 |  |  | 12
NYHA Functional Class [Count of Participants; unit: Participants] — Measure Description: NYHA Classification - The stages of heart failure: 1. Class I - No symptoms and no limitation in ordinary physical activity 2. Class II - Mild symptoms and slight limitation during ordinary activity. 3. Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity. Comfortable only at rest. 4. Class IV - Severe limitations. Experiences symptoms even while at rest
  Participants
    Class 1 | 0 |  |  | 0
    Class II | 5 |  |  | 5
    Class III | 6 |  |  | 6
    Class IV | 1 |  |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of MR ≤ 2+ and Hierarchical Comparison of Randomized Device and Randomized Control Groups [Cardiovascular Death, Number of Heart Failure Hospitalizations, Improvement in 6 MWT Distance (in Meters) and KCCQ (Number of Points Improved)].
Description: Hierarchical comparison of device and control groups (for randomized groups): MR ≤ 2+ and cardiovascular death, number of heart failure hospitalizations, improvement in 6 MWT distance (in meters) and KCCQ (number of points improved).
Time Frame: 1 year
Population: No patients were randomized, therefore no data was collected. This parameter is meant to be analyzed in hierarchical order for the randomized arms only.
Arm/Group | Experimental: Edwards Cardioband System | Control: No Intervention
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Number of Participants With Major Adverse Events (MAE) [Device Group Only]
Description: Overall rate of device and procedure related Major Adverse Events (MAEs) through 30 days post procedure (including death, stroke, myocardial infarction, pericardial effusion requiring drainage, left circumflex coronary artery injury requiring intervention, mitral valve reintervention, and access site and vascular complications requiring intervention
Time Frame: 30 days
Population: No patients were randomized, therefore no data was collected in the randomized phase.
Measure: Count of Participants; unit: Participants
Groups:
- Roll-in: Transcatheter mitral valve repair with the Edwards Cardioband System. This patient group is treated by physicians requiring additional training prior to beginning randomized cohort enrollment.
Arm/Group | Roll-in | Experimental: Edwards Cardioband System | Control: No Intervention
Number analyzed (Participants) | 8 | 0 | 0
Participants | 0 |  |

3. Secondary Outcome: Secondary Safety Endpoints [Device Group Only]
Description: Components will be calculated with 95% confidence intervals 1. Death 2. Stroke 3. Myocardial infarction 4. Pericardial effusion requiring drainage 5. Mitral valve reintervention 6. Access site and vascular complications requiring intervention 7. Left circumflex coronary artery injury requiring intervention 8. Need for a new permanent pacemaker
Time Frame: 30 days
Population: No patients were randomized, therefore no data was collected
Measure: Count of Participants; unit: Participants
Arm/Group | Roll-in | Experimental: Edwards Cardioband System | Control: No Intervention
Number analyzed (Participants) | 8 | 0 | 0
Participants | 0 |  |

4. Secondary Outcome: Secondary Endpoints Through 1 Year (Powered for Randomized Arms Only)
Description: The following key secondary efficacy endpoints will be tested in comparison to control in a hierarchical order to preserve statistical power. 1. MR ≤ 1+ 2. NYHA Class 3. Kansas City Cardiomyopathy Questionnaire (KCCQ) 4. 6 Minute Walk Test (6MWT) 5. SF-36v2 Health Survey (SF-36) 6. Heart Failure Hospitalizations 7. Cardiovascular mortality
Time Frame: 1 year
Population: No patients were randomized, therefore no data was collected. The parameter is meant to be analyzed in hierarchical order for the randomized arms only.
Arm/Group | Experimental: Edwards Cardioband System | Control: No Intervention
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Device Success
Description: Device is deployed as intended and the delivery system is successfully retrieved as intended at the time of the patient's exit from the cardiac catheterization laboratory (per device analysis).
Time Frame: 30 days
Population: No patients were randomized, therefore no data was collected in the randomized phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Roll-in | Experimental: Edwards Cardioband System | Control: No Intervention
Number analyzed (Participants) | 12 | 0 | 0
Participants | 8 |  |

6. Secondary Outcome: Procedural Success
Description: Device success with evidence of MR reduction to ≤ MR2+ at discharge and without the need for a surgical or percutaneous intervention prior to hospital discharge (per patient analysis).
Time Frame: 30 days
Population: No patients were randomized, therefore no data was collected in the randomized phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Roll-in | Experimental: Edwards Cardioband System | Control: No Intervention
Number analyzed (Participants) | 12 | 0 | 0
Participants | 7 |  |

7. Secondary Outcome: Clinical Success
Description: Procedural success with evidence of MR reduction ≤ MR2+ and without MAEs* at 30 days (per patient analysis). *Major adverse events (MAE) defined as death, stroke, myocardial infarction, pericardial effusion requiring drainage, left circumflex coronary artery injury requiring intervention, mitral valve reintervention and access site and vascular complications requiring intervention.
Time Frame: 30 days
Population: No patients were randomized, therefore no data was collected in the randomized phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Roll-in | Experimental: Edwards Cardioband System | Control: No Intervention
Number analyzed (Participants) | 12 | 0 | 0
Participants | 7 |  |

ADVERSE EVENTS:
Time Frame: 5 Years
Description: Trial was designed for patients to be randomized. No patients were randomized, therefore no data was collected for experimental or control groups
Arm/Group | Roll-in | Experimental: Edwards Cardioband System | Control: No Intervention
All-Cause Mortality (participants affected / at risk) | 4/12 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 9/12 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 8/12 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roll-in (N=12) | Experimental: Edwards Cardioband System (N=0) | Control: No Intervention (N=0)
Acute Left Ventricular Failure (Cardiac disorders) | 1 (1) | NA | NA
Atrial Fibrillation (Cardiac disorders) | 2 (2) | NA | NA
Atrial Flutter (Cardiac disorders) | 2 (3) | NA | NA
Cardiac Failure (Cardiac disorders) | 1 (2) | NA | NA
Cardiac Failure Acute (Cardiac disorders) | 2 (11) | NA | NA
Cardiac Failure Congestive (Cardiac disorders) | 2 (4) | NA | NA
Cardiogenic Shock (Cardiac disorders) | 1 (1) | NA | NA
Mitral Valve Incompetence (Cardiac disorders) | 1 (2) | NA | NA
Pericardial Effusion (Cardiac disorders) | 1 (1) | NA | NA
Pulmonary Oedema (Cardiac disorders) | 1 (1) | NA | NA
Death (General disorders) | 1 (1) | NA | NA
Clostridium Difficile Colitis (Infections and infestations) | 1 (1) | NA | NA
Sepsis (Infections and infestations) | 1 (1) | NA | NA
Septic Shock (Infections and infestations) | 1 (1) | NA | NA
Clavicle Fracture (Injury, poisoning and procedural complications) | 1 (1) | NA | NA
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | NA | NA
Dehydration (Metabolism and nutrition disorders) | 1 (1) | NA | NA
Gout (Metabolism and nutrition disorders) | 1 (1) | NA | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | NA | NA
Device Dislocation (Product Issues) | 1 (1) | NA | NA
Urinary Retention (Renal and urinary disorders) | 1 (1) | NA | NA
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (4) | NA | NA
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | NA
Hypotension (Vascular disorders) | 1 (1) | NA | NA
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | NA | NA
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | NA
Cardiac Resynchronisation Therapy (Surgical and medical procedures) | 1 (1) | NA | NA
Chronic Left Ventricular Failure (Cardiac disorders) | 1 (1) | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roll-in (N=12) | Experimental: Edwards Cardioband System (N=0) | Control: No Intervention (N=0)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | NA | NA
Atrial Fibrillation (Cardiac disorders) | 2 (2) | NA | NA
Atrioventricular Block First Degree (Cardiac disorders) | 1 (1) | NA | NA
Cardiac Failure (Cardiac disorders) | 1 (1) | NA | NA
Mitral Valve Incompetence (Cardiac disorders) | 1 (1) | NA | NA
Nodal Rhythm (Cardiac disorders) | 1 (1) | NA | NA
Supraventricular Extrasystoles (Cardiac disorders) | 1 (1) | NA | NA
Tricuspid Valve Incompetence (Cardiac disorders) | 1 (1) | NA | NA
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | NA | NA
Hypothyroidism (Endocrine disorders) | 1 (1) | NA | NA
Asthenia (General disorders) | 1 (1) | NA | NA
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | NA | NA
Humerus Fracture (Injury, poisoning and procedural complications) | 1 (1) | NA | NA
Medical Device Site Injury (Injury, poisoning and procedural complications) | 1 (1) | NA | NA
Electrocardiogram Qt Prolonged (Investigations) | 1 (1) | NA | NA
Troponin I Increased (Investigations) | 1 (1) | NA | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | NA | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (2) | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | NA | NA
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | NA | NA
Acute Kidney Injury (Renal and urinary disorders) | 2 (2) | NA | NA
Renal Impairment (Renal and urinary disorders) | 1 (1) | NA | NA
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | NA
Air Embolism (Vascular disorders) | 1 (1) | NA | NA
Haematoma (Vascular disorders) | 1 (1) | NA | NA
Hypotension (Vascular disorders) | 1 (1) | NA | NA
Bundle Branch Block Right (Cardiac disorders) | 1 (1) | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-04-20): https://cdn.clinicaltrials.gov/large-docs/75/NCT03016975/Prot_002.pdf
  • Statistical Analysis Plan (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/75/NCT03016975/SAP_003.pdf